CLINICAL TRIAL: NCT00140894
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Rofecoxib in Familial Adenomatous Polyposis (FAP)
Brief Title: A Study of Rofecoxib in Familial Adenomatous Polyposis (FAP) (0966-205)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-205; 2005_052
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Adenomatous Polyposis Coli
Keywords: Osteoarthritis; Cancer Pain
MeSH Terms: conditions — Adenomatous Polyposis Coli; Osteoarthritis; Cancer Pain | interventions — rofecoxib; Duration of Therapy

INTERVENTIONS:
Drug: MK0966; rofecoxib / Duration of Treatment: 24 weeks
Drug: Comparator: placebo / Duration of Treatment: 24 weeks

SUMMARY:
A study to evaluate rofecoxib in the treatment of rectal, colon, or duodenal adenomas in patients with Familial Adenomatous Polyposis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age with familial adenomatous polyposis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62
Dates: Start 2002-08-06 (Actual); Study Completion 2004-10-11 (Actual)

PRIMARY OUTCOMES:
Number and average size of rectal polyps
Safety and tolerability

SECONDARY OUTCOMES:
Number and average size of duodenal polyps
Proportions of patients with improved overall colon rating

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php